CLINICAL TRIAL: NCT05415033
Title: Validity and Reliability of Arabic Version of Breast Questionnaire for Post Mastectomy Patients
Brief Title: Validity and Reliability of Arabic Version of Breast Questionnaire
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, gehad emad el din abd elaziz dandash, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Arabic BREAST-Q
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: BREAST-Q

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BREAST-Q (Other)
  Interventions: Other: BREAST-Q

INTERVENTIONS:
Other: BREAST-Q — arabic version of breast questionnaire

SUMMARY:
To test validity and reliability of the translated Arabic version of breast questionnaire .

DETAILED DESCRIPTION:
Breast cancer is the second most common cancer among women in the United States, with an estimated 246,660 .

Breast cancer patients and survivors now have many surgical options, which emphasizes the importance of understanding the long-term quality of life (QOL) outcomes Women undergoing surgery for primary breast cancer are increasingly making their own surgical decisions, and are often choosing between breast conserving therapy and mastectomy with or without breast reconstruction Although recent studies suggest breast conserving therapy has a survival benefit patients often turn to satisfaction and QOL outcomes data to help guide the decision - making process .

In the treatment of the special type of breast cancer (STBC), the choice of chemotherapeutic agents is often based on the characteristic features of the histological type .

On the other hand, the surgical strategy is usually determined by the tumor size and presence of lymph node metastasis, and the indication for immediate reconstruction is rarely discussed based on the histological type .

A mastectomy is used to remove all breast tissue if you have breast cancer or are at very high risk of developing it. You may have a mastectomy to remove one breast (unilateral mastectomy) or both breasts (bilateral mastectomy) For those with early-stage breast cancer, there are two optiones a mastectomy and Breast-conserving surgery (lumpectomy), in which only the tumor is removed from the breast, may be another option .

Choosing between a mastectomy and lumpectomy can be difficult. Both procedures are equally effective for preventing a recurrence of breast cancer. But a lumpectomy isn't an option for everyone with breast cancer .

Newer mastectomy techniques can preserve breast skin and allow for a more natural breast appearance following the procedure. This is also known as skin- sparing mastectomy Surgery to restore shape to your breast - called breast reconstruction - may be done at the same time as your mastectomy or during a second operation at a later date .

The BREAST-Q can provide meaningful data that can be used to support quality metrics and evidence-guided surgical practices in oncologic breast and plastic surgery It has been widely used by clinicians and researchers to help patients and surgeons better understand outcomes .

Since BREAST-Q was developed in 2009, it has been widely used by clinicians and researchers to capture information regarding health-related quality of life (HRQoL) and patient satisfaction related to breast surgery .

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent to a mastectomy operation.
* Patients ages between 30 to 60 years.
* All participants able to read and write in Arabic.
* All participants can understand items of the questionnaire.

Exclusion Criteria:

* Patients with mental problems.
* Patient with communication, vision, hearing disorders.
* Patient who doesn't fill the questionnaire till the end.
* Patient who isn't cooperative in filling the questionnaire.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 87 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
SATISFACTION WITH BREASTS | 3 monthes
  With your breast area in mind, in the past week, how satisfied or dissatisfied have you been with

SECONDARY OUTCOMES:
PSYCHOSOCIAL WELL-BEING | 3 monthes
  With your breast area in mind, in the past week, how often have you felt

OTHER OUTCOMES:
SEXUAL WELL-BEING | 3 monthes
  Thinking of your sexuality, how often do you generally feel
PHYSICAL WELL-BEING: CHEST | 3 monthes
  In the past week, how often have you experienced
ADVERSE EFFECTS OF RADIATION | 3 monthes
  If you have had radiation on both breasts, answer these questions thinking of the breast you are least satisfied with. With your radiated breast(s) in mind, in the past week, how much have you been bothered
CANCER WORRY | 3 monthes
  These statements ask about the WORRY you may be experiencing about breast cancer
FATIGUE | 3 monthes
  Does FATIGUE (feeling tired) from breast cancer or its treatment affect your quality of life?
IMPACT ON WORK | 3 monthes
  Does breast cancer or its treatment affect your WORK LIFE? Please answer thinking of when you were last working.
SATISFACTION WITH MEDICAL TEAM | 3 monthes
  These questions ask about your breast cancer surgeon , members of the medical team other than the surgeon, members of the office staf